CLINICAL TRIAL: NCT05789056
Title: A Multicenter, Open Label Study of QRX003 Lotion in Subjects With Netherton Syndrome
Brief Title: Open Label, Safety and Efficacy Study of QRX003 Lotion in Subjects With Netherton Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Quoin Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-QRX003-002
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Intervention Model Description: Open Label
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- QRX003, 4% QAM (Experimental): Subjects will apply test article once daily in the morning (QAM) for 12 weeks
  Interventions: Drug: QRX003, 4% Lotion
- QRX003, 4% BID (Experimental): Subjects will apply test article twice daily (BID) for 12 weeks
  Interventions: Drug: QRX003, 4% Lotion

INTERVENTIONS:
Drug: QRX003, 4% Lotion — QRX003Topical Lotion containing 4% active drug (serine protease inhibitor)

SUMMARY:
To assess the safety, tolerability, and efficacy of QRX003 lotion (4%) when added to standard of care treatment regimen, including systemic therapy in subjects with Netherton syndrome

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female at least 14 years of age.
* Females must be post-menopausal , surgically sterile , or use an effective method of birth control , for the duration of the study and for 3 months following completion of treatment. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Screening and Visit 2/Baseline.
* Subject has a clinical diagnosis of NS and agrees to genetic testing at Visit 1/Screening for confirmation of NS diagnosis if the subject does not have test results confirming a SPINK5 mutation.
* Subject has NS lesions in the Treatment Area (i.e., arms or lower legs).
* Subject is in good general health and free of any disease state or physical condition that might impair evaluation of NS or exposes the subject to an unacceptable risk by study participation.
* Subject is on a stable treatment regimen including systemic therapy for NS prior to baseline that is expected to remain stable for the duration of the study

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has any skin pathology in the Treatment Area or condition that, could interfere with the evaluation of the test article or requires use of interfering topical, systemic, or surgical therapy.
* Subject has active cancer of any type excluding non-melanoma skin cancer outside of the Treatment Area.
* Subject has diabetes of any type, except non-insulin dependent diabetes mellitus that is reasonably controlled.
* Subject has evidence of active infection during screening, or serious infection within 30 days prior to Visit 2/Baseline.
* Subject has known human immunodeficiency virus, hepatitis B or C virus, or active or latent tuberculosis.
* Subject has used ultraviolet phototherapy within the Treatment Area within 4 weeks prior to Visit 2/Baseline.
* Subject has used topical prescription treatment in the Treatment Area within 2 weeks prior to Visit 2/Baseline.
* Subject has used any topical bland moisturizers/emollients in the Treatment Area within 24 hours prior to Visit 2/Baseline.
* Subject is currently enrolled in an investigational drug, biologic, or device study.
* Subject has used an investigational drug, biologic, or device treatment within 30 days prior to Visit 2/Baseline.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with 1-point reduction on IGA | Up to week 16
  Proportion of subjects with 1-point reduction on the Investigator's Global Assessment (IGA) from Baseline. The IGA assesses overall severity of a subject's NS based on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Proportion of subjects with 2-point reduction on IGA | Up to week 16
  Proportion of subjects with 2-point reduction in IGA from Baseline.
NS surface area change | Up to week 16
  Change from Baseline in total Body Surface Area (BSA) affected by NS in the Treatment Area
WI-NRS score change | Up to week 16
  Change from Baseline in the Worst Itch-Numeric Rating Scale (WI-NRS) score ≥4. Itch severity is graded on an 11-point scale where 0 represents "no itch" and 10 represents "worst itch imaginable".
Assessment of subject satisfaction with treatment based on TSQM | Up to week 16
  Assessment of subject satisfaction with treatment based on the Treatment Satisfaction Questionnaire for Medication (TSQM). The TSQM measures a subject's level of satisfaction or dissatisfaction with the treatment. Composite scores can range from 0 to 100; higher scores indicate better satisfaction.
Proportion of subjects requiring rescue therapy | Up to week 16
  Proportion of subjects requiring rescue therapy
Safety Assessment-AEs | Up to week 16
  Any local and systemic AEs (Adverse Events)/serious AEs
Safety Assessment-LSRs | Up to week 16
  Number of subjects with presence of the following LSRs (Local Skin Reactions): edema, excoriations, oozing/vesiculation/crusting, and erosions at any study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Andrasfay, Study Director — Therapeutics, Inc.
Locations (4):
- United States (4):
  - Site #1, San Diego, California
  - Site #4, Indianapolis, Indiana
  - Site #5, Quincy, Massachusetts
  - Site #2, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No